CLINICAL TRIAL: NCT01926613
Title: Cognitive Rehabilitation and Supported Employment for Severe Mental Illness
Brief Title: Thinking Skills for Work in Severe Mental Illness
Acronym: TSW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH077210; 1R01MH077210-01 (NIH)
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Major Depression; Bipolar Disorder; Anxiety Disorder
Keywords: Schizophrenia; Chronic Mental Disorder; Employment; Cognitive remediation; Vocational rehabilitation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Depressive Disorder, Major; Bipolar Disorder; Anxiety Disorders | interventions — Employment, Supported

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supported Employment Only (Active Comparator): Supported employment is an evidence based practice designed to help people with serious mental illness obtain competitive work. This vocational model adheres to the principles of zero inclusion, rapid job search, no prevocational training, attention to client preferences and integration with clinical services.
  Interventions: Behavioral: Supported Employment
- Thinking Skills for Work (Experimental): The Thinking Skills for Work Program includes 5 components delivered by a Cognitive Specialist who works collaboratively with the consumer's Employment Specialist: a) assessing the consumer's strengths and weaknesses in cognitive functioning, and analysis of the contribution of cognitive impairments and other factors to job losses and difficulties obtaining a job; b) teaching coping strategies for dealing with cognitive challenges associated with job search or maintaining a job; c) computer cognitive training involving cognitive exercises with a commercially available software program, which is designed to improve the broad range of cognitive skills through a combination of practice and strategy coaching by the Cognitive Specialist; d) job search planning; and e) job support consultation.
  Interventions: Behavioral: Thinking Skills for Work Program

INTERVENTIONS:
Behavioral: Thinking Skills for Work Program — The Thinking Skills for Work includes assessment of cognitive strengths and weaknesses and their relationship with work history, computerized cognitive practice, compensatory strategy training, and integration of cognitive and supported employment services.
  Arms: Thinking Skills for Work
Behavioral: Supported Employment — Supported Employment is an evidence based vocational rehabilitation program
  Arms: Supported Employment Only

SUMMARY:
The purpose of this study is help people with serious mental illness and receiving vocational rehabilitation get and keep the job they want by improving their thinking skills, such as attention and memory, using computer exercises and other strategies. One half of the participants in the study will receive vocational rehabilitation and the exercises to improve thinking skills, and the other half will receive just vocational rehabilitation. All participants will receive an assessment of symptoms and thinking skills at the beginning of the study and 6, 12, and 24 months later. Work activity during the 24 months in the study will be collected. It is expected that those participants who receive the practice of their thinking skills will be more likely to get and keep the job they want compared with people who do not receive this treatment.

DETAILED DESCRIPTION:
This randomized controlled trial is evaluating the effectiveness of a pilot-tested, manualized cognitive remediation intervention entitled the "Thinking Skills for Work Program" by comparing it to enhanced supported employment services in clients with severe mental illness (SMI) who are participants in high fidelity supported employment programs at the Greater Mental health Center of Manchester and Thresholds, Inc., Chicago, Il, but who have had difficulty getting or keeping jobs. Participants are randomized to either the Thinking Skills for Work (cognitive remediation +supported employment; CT+SE) or enhanced supported employment (E-SE), with cognitive, symptom, and quality of life assessments performed at baseline, 3 months (following the completion of the computerized cognitive training component of the Thinking Skills for Work program), 12 months, and 24 months, and employment data gathered over the full 2-year period. For the E-SE condition, supported employment services are enhanced by training provided to the employment specialists regarding to recognize cognitive problems related to work performance, and how employment specialists can teach clients coping strategies for managing these problems. Primary analyses will focus on testing the hypotheses that the Thinking Skills for Work Program (CT+SE) leads to better cognitive functioning and better competitive work outcomes over the 2-year follow-up period compared to the E-SE program.

ELIGIBILITY:
Inclusion Criteria:

* Chronic mental disorder
* Minimum age 18
* Unemployed
* Wants employment
* Must be a recipient of services at one of two participating agencies
* Fluent in English
* Willing and legally able to provide informed consent to participate in study -Subjects with court appointed legal guardians will be included

Exclusion Criteria:

* History of neurological conditions that impair cognition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2006-04; Primary Completion 2009-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
AMOUNT OF EMPLOYMENT | 24 months
  TOTAL HOURS OF COMPETITIVE EMPLOYMENT FROM BASELINE TO 24 MONTHS. TOTAL WEEKS OF EMPLOYMENT FROM BASELINE TO 24 MONTHS. TOTAL NUMBER OF JOBS HELD FROM BASELINE TO 24 MONTHS.

SECONDARY OUTCOMES:
EXECUTIVE FUNCTIONING AND MEMORY | BASELINE, 6, 12, and 24 months
  CHANGE FROM BASELINE IN EXECUTIVE FUNCTIONING AND MEMORY AT 6 MONTHS USING THE MATRICS COGNITIVE ASSESSMENT BATTERY. CHANGE FROM BASELINE IN EXECUTIVE FUNCTIONING AND MEMORY AT 12 MONTHS USING THE MATRICS COGNITIVE ASSESSMENT BATTERY.. CHANGE FROM BASELINE IN EXECUTIVE FUNCTIONING AND MEMORY AT 24 MONTHS USING THE MATRICS COGNITIVE ASSESSMENT BATTERY.

CONTACTS AND LOCATIONS:
Overall Officials: Susan R McGurk, Ph.D., Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (2):
- United States (2):
  - Thresholds, Inc., Chicago, Illinois
  - Mental Health Center of Greater Manchester, Manchester, New Hampshire

REFERENCES:
- [Derived] McGurk SR, Mueser KT, Xie H, Welsh J, Kaiser S, Drake RE, Becker DR, Bailey E, Fraser G, Wolfe R, McHugo GJ. Cognitive Enhancement Treatment for People With Mental Illness Who Do Not Respond to Supported Employment: A Randomized Controlled Trial. Am J Psychiatry. 2015 Sep 1;172(9):852-61. doi: 10.1176/appi.ajp.2015.14030374. Epub 2015 May 22. PMID 25998278